CLINICAL TRIAL: NCT03081624
Title: Evaluation of Neurological Status and School Readiness of Preterm Children in Preschool Period
Brief Title: Evaluation of Neurological Status and School Readiness in Preterm Preschoolers
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Ramazan Yildiz, Research Assistant, Gazi University
Other Study IDs: E.5461
Record Dates: First submitted 2017-03-10; First posted 2017-03-16 (Actual); Last update posted 2017-04-25 (Actual); Status verified 2017-03

CONDITIONS: School Readiness
Keywords: preterm; neurological status; School Readiness
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Preterm Preschoolers: Preterm children who haven't attend school.
- Term Preschoolers: Term children who haven't attend school.

SUMMARY:
Beginning school is an important milestone for children. Children's readiness for school involves cognitive, physical, and emotional development. While the majority of children born preterm are able to transition from preschool to kindergarten with little difficulty, some children experience challenges during this time. Factors that negatively influence children's success in kindergarten include their age, socioeconomic status, neurological status and their ability to interpret sensory information from their environment.

This study was planned to explain the relationship between the primary school readiness and the neurological status of preterm born children.

DETAILED DESCRIPTION:
A convenience of preterm and term preschoolers recruiting from Gazi University, Faculty of Health Science, Department of Physiotherapy and Rehabilitation. Each group contains 30 children. First, sociodemographic information and histories of children are obtaining. Ages and contact information of the parents are recording. Prenatal and natal risk factors of the mothers are querying. Gestational ages and height, weight, and head circumferences of babies at birth are recording. Number of pregnancies, live births and abortions, type of delivery, multiple pregnancies for mothers as well as consanguinity between parents are asking. Marmara Primary School Readiness Scale is using to evaluate mental-language development, socio-emotional development, physical development, self-care skills,math skills, science skills, voice exercises, line exercises and labyrinths. Sensory profile caregiver questionnaire screen for the senses (sensory processing), adjustment (modulation), behavioral and emotional responses. The Touwen examination (neurological examination) is using to evaluate posture in various positions, muscle tone, dyskinesias, range of motion, reflexes, sensory function and cranial nerve function as well as developmental items, i.e. the items dealing with coordination, fine manipulative abilities and associated movements. All examination wiil be finished in the same day.

ELIGIBILITY:
Inclusion Criteria:

* No neurological diagnosis
* gestational age < 37 weeks
* 60-78 months of age

Exclusion Criteria:

* Have a neurological diagnosis (such as cerebral palsy)
* Grade III or grade IV intraventricular hemorrhage
* Have undergone major surgery in neonatal period
* Mental retardation

Ages: 60 Months to 78 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Preterm children and their age -matched term volunteers
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2016-12-17 (Actual); Primary Completion 2017-07-17 (Estimated); Study Completion 2018-07-17 (Estimated)

PRIMARY OUTCOMES:
Marmara Primary School Readiness Scale | 45 minutes
  The application form includes math skills, science skills, voice exercises, line exercises and labyrinths; Development form; Mental-language development, socio-emotional development, physical development, self-care skills.

SECONDARY OUTCOMES:
Sensory profile caregiver questionnaire | 45 minutes
  The profile reveals the child's sensory appearance in terms of sensory search, emotional response formation, low endurance, oral tenderness, distractibility, weak perception, sensory sensitivity, activity level and fine motor / perceptual differences. In addition, the child evaluates the senses (sensory processing), adjustment (modulation), behavioral and emotional responses.
The Touwen examination (neurological examination) | 45 minutes
  The assesment includes traditional neurological items, such as the evaluation of posture in various positions, muscle tone, dyskinesias, range of motion, reflexes, sensory function and cranial nerve function as well as developmental items, i.e. the items dealing with coordination, fine manipulative abilities and associated movements.

CONTACTS AND LOCATIONS:
Overall Officials: Bülent Elbasan, Phd, Study Chair — Gazi University

IPD SHARING:
Plan to Share IPD: Undecided
Haven't decided yet.